CLINICAL TRIAL: NCT00612768
Title: Clinical Evaluation of T.R.U.E. TEST® Fragrance Mix and Thimerosal Allergens: Bioequivalence of Polyvinylpyrrolidone (PVP) Formulations
Brief Title: Clinical Evaluation of T.R.U.E. TEST® Fragrance Mix and Thimerosal Allergens:Bioequivalence of PVP Formulations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allerderm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Mekos 07 2P1/2 401; 20071738 (Other: Western Institutional Review Board)
Record Dates: First submitted 2008-01-30; First posted 2008-02-12 (Estimated); Results first posted 2018-04-09 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Dermatitis, Contact
Keywords: Bioequivalence; Thimerosal; Fragrance Mix; PVP formulation; Contact dermatitis
MeSH Terms: conditions — Dermatitis, Contact | interventions — Thimerosal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- T.R.U.E. Test allergens Fragrance Mix and Thimerosol (Experimental): Concordance (agreement) between positive patch reactions to
  1. fragrance mix (0.43 mg/cm2) in polyvinylpyrrolidone (PVP) vs fragrance mix (0.43 mg/cm2) in hydroxypropylcellulose (HPC)
  2. thimerosol (0.008 mg/cm2) in polyvinylpyrrolidone (PVP) vs thimerosol (0.008 mg/cm2) in hydroxypropylcellulose (HPC)
  3. fragrance mix T.R.U.E. Test allergen vs fragrance mix reference allergen (petrolatum)
  4. thimerosol T.R.U.E. Test allergen vs thimerosol reference allergen (petrolatum)
  will be measured
  Interventions: Biological: TRUE Test allergens Fragrance Mix and Thimerosol

INTERVENTIONS:
Biological: TRUE Test allergens Fragrance Mix and Thimerosol — * Thimerosal, 0.008 mg/cm2 in hydroxypropylcellulose
  * Thimerosal, 0.008 mg/cm2 in polyvinylpyrrolidone
  * Fragrance mix, 0.43 mg/cm2 in hydroxypropylcellulose with β-cyclodextrin
  * Fragrance mix, 0.43 mg/cm2 in polyvinylpyrrolidone with β-cyclodextrin
  Patches are placed at day one and removed 48 hours. The duration of the study lasts 21 days. However, the subject is only exposed the the study allergen for 48 hours.
  Other Names: T.R.U.E. TEST Skin Patch Test

SUMMARY:
Open, prospective, multi-center study to evaluate the bioequivalence of povidone (PVP) formulations of 2 T.R.U.E. TEST allergens: fragrance mix and thimerosal.

DETAILED DESCRIPTION:
Bioequivalence will be determined in 40 adult subjects (20 per allergen), who have a clinical history of contact dermatitis and have tested positive to fragrance mix or thimerosal.

ELIGIBILITY:
Inclusion Criteria:

* Current or previous symptoms and/or history consistent with allergic contact dermatitis, and positive patch test (within the past 5 years) to fragrance mix AND/OR thimerosal.
* All subjects must be adults (18 years of age or older) and otherwise in good health.
* Pre-menopausal female subjects must consent to a urine pregnancy test; results must be negative for study inclusion.
* Informed consent must be signed and understood by each subject, and consistent with all institutional, local and national regulations.

Exclusion Criteria:

* Subjects unable to meet inclusion requirements.
* Women who are breastfeeding or pregnant.
* Topical treatment during the last 7 days with corticosteroids or other immunosuppressive agents on or near the test area.
* Systemic treatment during the last 7 days with corticosteroids (equivalent to > 10 mg prednisone) or other immunosuppressive agents.
* Treatment with ultraviolet (UV) light (including tanning) during the previous 3 weeks.
* Acute dermatitis outbreak or dermatitis on or near the test area on the back.
* Subjects unable to comply with patch test study requirements including multiple return visits and activity restrictions (e.g., protecting test panels from excess moisture due to showering or vigorous activity).
* Subject participation in clinical trials of investigational drugs, treatments, or devices, other than T.R.U.E. TEST, during this study or 3 weeks prior to inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Fowler, MD, Principal Investigator — Dermatology Specialists PSC; Luz Fonacier, MD, Principal Investigator — Winthrop University Hospital; Donald V. Belsito, MD, Principal Investigator — American Dermatology Associates; Jerri Hoskyn, MD, Principal Investigator — River City Dermatology
Locations (4):
- United States (4):
  - River City Dermatology, Little Rock, Arkansas
  - American Dermatology Associates, Shawnee Mission, Kansas
  - Dermatology Specialists PSC, Louisville, Kentucky
  - Winthrop University Hospital, Mineola, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 4 centers in the United States. The first subject was enrolled on Jan 2 2008 and the study completed on Dec 12 2008.
Pre-assignment Details: No subject was excluded from the trial following enrollment but before assignment to a group.
Groups:
- Sensitive Subjects: All subjects recruited to this study were to have had previous positive patch test results to one of the allergens tested on the study.
Period: Overall Study
Arm/Group | Sensitive Subjects
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Sensitive Subjects: Subjects with a clinical history and positive patch test (current or previous) to either fragrance mix or thimerosal. Study subjects must be otherwise healthy and fulfill entry criteria.
Arm/Group | Sensitive Subjects
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (16.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Analysis of Bioequivalence: Concordance
Description: Percent agreement between T.R.U.E. Test allergen in PVP vs HPC is based on a positive test response during at least one post application visit
Time Frame: Up to 21 days
Population: The data from 50 subjects enrolled in the study was analyzed
Measure: Number (95% Confidence Interval); unit: percentage of agreement
Groups:
- Fragrance Mix; Thimerosol: Percent agreement between T.R.U.E. Test allergen in PVP vs HPC
Arm/Group | Fragrance Mix | Thimerosol
Number analyzed (Participants) | 50 | 50
percentage of agreement | 76 [61.8 to 86.9] | 98.0 [89.4 to 99.9]

2. Primary Outcome: Agreement Between TRUE Test Allergen and Reference Allergen
Description: Sensitivity: Agreement between positive results for the test and reference allergen Specificity: Agreement between negative results for the test and reference allergen
Time Frame: Up to 21 days
Population: The data from all enrolled subjects was analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of agreement
Groups:
- Sensitivity: Fragrance Mix in HPC; Sensitivity: Fragrance Mix in PVP; Sensitivity: Thimerosal in HPC; Sensitivity: Thimerosol in PVP: Agreement between positive results for the test and reference allergen
- Specificity: Fragrance Mix in HPC; Specificity: Fragrance Mix in PVP; Specificity: Thimerosal in HPC; Specificity: Thimerosal in PVP: Agreement between negative results for the test and reference allergen
Arm/Group | Sensitivity: Fragrance Mix in HPC | Sensitivity: Fragrance Mix in PVP | Sensitivity: Thimerosal in HPC | Sensitivity: Thimerosol in PVP | Specificity: Fragrance Mix in HPC | Specificity: Fragrance Mix in PVP | Specificity: Thimerosal in HPC | Specificity: Thimerosal in PVP
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 50 | 50 | 50
percentage of agreement | 40.9 [20.7 to 63.6] | 59.1 [36.4 to 79.3] | 61.5 [40.6 to 79.8] | 65.4 [44.3 to 82.8] | 92.9 [76.5 to 99.1] | 100 [87.7 to 100] | 100 [85.8 to 100] | 100 [85.8 to 100]

3. Secondary Outcome: Irritation, Adhesion, Itching/Burning
Description: Frequency of tape-induced irritation at the test site, incomplete panel adhesion and subject-reported sensations of itching or burning.
Time Frame: Visit 2: 48 hours after patch application
Measure: Number; unit: percentage of participants
Groups:
- Tape Irritation: TRUE Test Panel: Percentage of participants who exhibited tape-induced irritation at visit 2.
- Incomplete Panel Adhesion: TRUE Test; Incomplete Panel Adhesion: Reference Allergen: Percentage of participants whose panels were not 100% adhered at visit 2.
- Itching and Burning: Percentage of participants who reported patch related itching and/or burning at visit 2
Arm/Group | Tape Irritation: TRUE Test Panel | Incomplete Panel Adhesion: TRUE Test | Incomplete Panel Adhesion: Reference Allergen | Itching and Burning
Number analyzed (Participants) | 50 | 50 | 50 | 50
percentage of participants | 28 | 24 | 20 | 46

4. Secondary Outcome: Frequency of Late and Persistent Reactions
Description: Late reactions occur 7-10 days after patch application Persistent reactions initially occur at 2-4 days after application and persist through 7-21 days after application
Time Frame: Day 2 (48 hours after application) through Day 21
Measure: Number; unit: percentage of subjects with reactions
Groups:
- Late Reactions: Fragrance Mix in HPC; Late Reactions: Fragrance Mix in PVP; Late Reactions: Thimerosal in HPC; Late Reactions: Thimerosol in PVP: Late reactions occur 7-10 days after patch application
- Persistent Reactions: Fragrance Mix in HPC; Persistent Reactions: Fragrance Mix in PVP; Persistent Reactions: Thimerosal in HPC; Persistent Reactions: Thimerosal in PVP: Persistent reactions initially occur at 2-4 days after application and persist through 7-21 days after application
Arm/Group | Late Reactions: Fragrance Mix in HPC | Late Reactions: Fragrance Mix in PVP | Late Reactions: Thimerosal in HPC | Late Reactions: Thimerosol in PVP | Persistent Reactions: Fragrance Mix in HPC | Persistent Reactions: Fragrance Mix in PVP | Persistent Reactions: Thimerosal in HPC | Persistent Reactions: Thimerosal in PVP
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 50 | 50 | 50
percentage of subjects with reactions | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4

ADVERSE EVENTS:
Time Frame: Day 0-21
Groups:
- Sensitives: subjects per allergen with a clinical history and positive patch test (current or previous) to either fragrance mix or thimerosal. Study subjects must be otherwise healthy and fulfill entry criteria.
Arm/Group | Sensitives
Serious Adverse Events (participants affected / at risk) | 1/50
Other Adverse Events (participants affected / at risk) | 5/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sensitives (N=50)
Right femoral sheath placed secondary to tronsientischemic attack/carotid stenosis (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sensitives (N=50)
Bladder Infection (Gastrointestinal disorders) | 1
Itching (Skin and subcutaneous tissue disorders) | 1
Itching and burning (Skin and subcutaneous tissue disorders) | 1
Itching on/around site (Skin and subcutaneous tissue disorders) | 1
Reports burning sensation, she thinks it might be due to the tape (Skin and subcutaneous tissue disorders) | 1
Itching at positive patch sites (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No